CLINICAL TRIAL: NCT03139214
Title: Parenting Intervention and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000856
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention involved 7 parenting sessions with mothers and their children that taught nurturant parenting techniques, effective communication skills, and about the importance of developing and following household rules.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parenting intervention, 7 weekly sessions, each session 2 hours in length.
  Interventions: Behavioral: Parenting Intervention
- Control (No Intervention): 3 mailings about child development and stress management.

INTERVENTIONS:
Behavioral: Parenting Intervention
  Arms: Intervention

SUMMARY:
This study aimed to test the effect of a parenting intervention on metabolic syndrome in African American youth. The investigators hypothesized that a parenting intervention would produce reductions in metabolic syndrome, particularly for those families that started out high in difficulties with parenting.

DETAILED DESCRIPTION:
In this study, the investigators conducted a parenting intervention (Strong African American Families, or SAAF). Families (mothers with their 11 year old child) were randomized to either the parenting intervention or to a control group. Those in the intervention group received 7 group sessions with the parent and child aimed at promoting better family relationships. Those in the control group received 3 mailings about child development and stress management. At age 25, youth were assessed on metabolic syndrome. The investigators hypothesized that the parenting intervention would produce reductions in metabolic syndrome relative to the control group, particularly for those families that started out high in difficulties with parenting.

ELIGIBILITY:
Inclusion Criteria: 5th graders -

Exclusion Criteria: None

-

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 391 (Actual)
Dates: Start 2001-08-27 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome diagnosis (based on International Diabetes Federation criteria using a clinical assessment of obesity, blood pressure, cholesterol, glucose) | 14 years post-intervention
  Metabolic syndrome diagnosis
Metabolic syndrome components | 14 years post-intervention
  Number of components of metabolic syndrome that were clinically elevated

IPD SHARING:
Plan to Share IPD: No